CLINICAL TRIAL: NCT02328183
Title: Efficacy of Polymyxin B Against Infections Caused by Extensively Drug-resistant (XDR) Gram-Negative Bacteria
Acronym: XDR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 568/2557(EC4)
Record Dates: First submitted 2014-12-15; First posted 2014-12-31 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Hospital Infection
Keywords: polymyxin B; carbapenem resistant bacteria
MeSH Terms: conditions — Cross Infection | interventions — Polymyxin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polymyxin B (Experimental): Polymyxin B 1.5-2.5 mg/kg/day intravenous q 12 hrs duration 7-14 days
  Interventions: Drug: Polymyxin B

INTERVENTIONS:
Drug: Polymyxin B — administrate drug by 0.75-1.25 mg/kg/dose intravenously q 12 hrs both saline and dextrose solution can be dissolved duration 7-14 days
  Other Names: X-Gen Phamaceuticals, USA Polymyxin B

SUMMARY:
The objective of the study is to evaluate the efficacy of Polymyxin B for treatment Gram negative bacterial infection. The hypothesis of study is Polymyxin B would be the new antibacterial agents for Thai Gram negative infected patients in case of desirable outcomes and minimal side effects.

DETAILED DESCRIPTION:
* Investigator is notified by doctors who take care of gram negative infected patients.
* Investigator inform patient or their relatives about all topics in project, eligible criteria, method, material and monitoring treatment.
* After patient or their relatives are appreciated to join this project, investigator collect data in case record form;electronics form, then implement the drug.
* Duration of treatment is determined by site and severity of infection, approximately 7-14 days.
* Sample size calculation, by prevalence formula, we estimate the mortality rate about 50 %, deviation 10 %,and 2-sided 95% Confidence interval, therefore,97 persons
* We estimate gather data about 100 persons.
* Statistical descriptive analysis for descriptive data.
* During the study is performing, all unexpected adverse event definitely report to Siriraj institutional Review Board immediately, in addition to subjects or their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 year-old
* The infection caused by carbapenem-resistant (CR) Enterobacteriaceae, CR P.aeruginosa or CR A. baumannii which susceptible to colistin
* The duration of treatment approximately between 7-14 days
* Kidney function, according to Kidney Disease Improving Global Outcomes (KDIGO) classification, should less than stage 4 and no replacement therapy in all modality.
* The patients are anticipated to live more than 48 hrs after participation.
* In case of Colistin administration beforehand, it should not exceed 24 hrs.
* All of participants should be willing to join this project.

Exclusion Criteria:

* Pregnancy and lactation
* End stage renal disease who take renal replacement therapy
* Any type of Neuromuscular disease
* Body mass index exceed 30
* Infection that require treatment more than 14 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
mortality rate | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  mortality rate of gram negative bacteria infected patients receiving Polymyxin B at day 28 after enrollment

SECONDARY OUTCOMES:
adverse drug reactions | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  we assess adverse drug reactions in 2 aspects; nephrotoxicity and neurotoxicity
microbiological clearance | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  we perform culture and staining to assess bacterial clearance after apply the study drug every 3 days until culture is negative
Peak Plasma Concentration (Cmax) of polymyxin B | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  we do the blood test for drug level at before the third date dose then 1,2,4 hours after administration of the polymixin B and before the fourth dose.

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Infectious disease and tropical medicine, Siriraj hospital
Locations (1):
- Siriraj hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Koomanachai P, Tiengrim S, Kiratisin P, Thamlikitkul V. Efficacy and safety of colistin (colistimethate sodium) for therapy of infections caused by multidrug-resistant Pseudomonas aeruginosa and Acinetobacter baumannii in Siriraj Hospital, Bangkok, Thailand. Int J Infect Dis. 2007 Sep;11(5):402-6. doi: 10.1016/j.ijid.2006.09.011. Epub 2007 Feb 8. PMID 17291803
- [Result] Nation RL, Velkov T, Li J. Colistin and polymyxin B: peas in a pod, or chalk and cheese? Clin Infect Dis. 2014 Jul 1;59(1):88-94. doi: 10.1093/cid/ciu213. Epub 2014 Apr 3. PMID 24700659